CLINICAL TRIAL: NCT04630639
Title: Validation of the Sparkle Respiratory Effort Signal Against Esophageal Pressure in Healthy Participants
Brief Title: Sparkle Respiratory Effort Validation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Changed scientific strategy. No participants were enrolled.
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Collaborators: Pulmonary Critical Care Associates of Baltimore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SRC-NBS-Sparkle-EP-2019-10456
Record Dates: First submitted 2020-11-09; First posted 2020-11-16 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Sleep Apnea, Obstructive; Sleep Apnea, Central
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea, Central

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Validation Arm (Experimental): Participants will wear the Sparkle device (test device) while instrumented with an esophageal manometry catheter (reference standard) to record respiratory effort.
  Interventions: Device: Sparkle

INTERVENTIONS:
Device: Sparkle — The Sparkle device is a single-use device intended to aid the diagnosis of sleep-disordered breathing; however, this study is intended only to validate the respiratory effort signal and does not assess diagnostic performance.

SUMMARY:
This study has been developed in order to demonstrate the validity of the Sparkle respiratory effort signal.

DETAILED DESCRIPTION:
The rationale for undertaking this study is to demonstrate that the agreement between the Sparkle respiratory effort signal amplitude and esophageal manometry is non-inferior to the agreement between the thoracic belt respiratory effort signal amplitude and esophageal manometry. Data collection will be completed within a single visit, in which participants will undergo simultaneous measurement using the Sparkle device, respiratory belts, and esophageal manometry. Data collection will be completed during wakefulness, while participants undergo a series of breathing maneuvers.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years;
* Fluent in English;
* Able to provide informed consent.

Exclusion Criteria:

* Contraindication to esophageal pressure monitoring, including a sensitive gag reflex (determined by a positive response to the screening question "do you sometimes or often gag while brushing your teeth?"), dysphagia, nasal obstruction, and/or esophageal disorder likely to impact placement of the balloon;
* History of allergic reactions to medical adhesives;
* Known allergy to lidocaine;
* Known seizure disorder;
* Severe medical condition (controlled or uncontrolled) impacting breathing including neuromuscular disease, chronic obstructive pulmonary disease, respiratory failure or insufficiency, or requirement for oxygen therapy;
* Chronic cardiopulmonary or renal disease, including a history of irregular heart rhythms;
* At risk for excessive bleeding including use of anticoagulants;
* An employee, or spouse of an employee, of a company that designs, sells, or manufactures sleep related products (including Philips);
* An employee, or spouse of an employee, of Pulmonary and Critical Care Associates of Baltimore.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Breath amplitude correlation | Baseline
  The primary endpoint is the average correlation co-efficient of the breath amplitude sequences extracted from the Sparkle and esophageal manometry respiratory effort signals, with respect to the average correlation co-efficient of the breath amplitude sequences extracted from the thoracic belt and esophageal manometry respiratory effort signals.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Schwartz, MD, Principal Investigator — Pulmonary and Critical Care Associates of Baltimore
Locations (1):
- Pulmonary and Critical Care Associates of Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No